CLINICAL TRIAL: NCT07403006
Title: Impact of Root Surface Conditioning With Erythritol Air Polishing Versus Hand Instrumentation on Recession Coverage Using the Modified Tunnel Technique and Subepithelial Connective Tissue Graft: A Randomized Clinical Trial
Brief Title: Impact of Root Surface Conditioning With Erythritol Air Polishing and Hand Instrumentation on Recession Coverage Using the Modified Tunnel Technique and Subepithelial Connective Tissue Graft.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WUM.Perio.06
Record Dates: First submitted 2026-01-21; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythritol Air-Polishing (Experimental): Sites with gingival recessions treated with root surface preparation using erythritol air-polishing prior to modified tunnel technique with subepithelial connective tissue graft.
  Interventions: Procedure: Erythritol Air-Polishing
- Manual Root Instrumentation (Active Comparator): Sites with gingival recessions treated with root surface preparation using manual Gracey curettes prior to modified tunnel technique with subepithelial connective tissue graft.
  Interventions: Procedure: Manual Root Instrumentation

INTERVENTIONS:
Procedure: Erythritol Air-Polishing — Root surface preparation performed using erythritol powder air-polishing (EMS AIRFLOW PLUS) prior to root coverage surgery with a modified tunnel technique and subepithelial connective tissue graft.
  Arms: Erythritol Air-Polishing
Procedure: Manual Root Instrumentation — Mechanical root surface preparation performed using manual Gracey curettes before root coverage surgery with a modified tunnel technique and subepithelial connective tissue graft.
  Arms: Manual Root Instrumentation

SUMMARY:
This study aims to evaluate whether the method of root surface preparation influences surgical outcomes. It will assess whether manual root instrumentation can be replaced by a less invasive erythritol air-polishing technique.

ELIGIBILITY:
Inclusion Criteria:

* Multiple RT1 and/or RT2 gingival recessions (Cairo 2011), symmetrical and bilateral, with a minimum height of ≥ 1 mm
* Full-mouth plaque score (FMPS) < 15% (assessed on four surfaces per tooth)
* Full-mouth bleeding on probing (FMBOP) < 15% (assessed on four surfaces per tooth)
* Detectable cemento-enamel junction (CEJ)
* Age ≥ 18 years

Exclusion Criteria:

* RT3 gingival recessions (Cairo 2011)
* Gingival recessions affecting second and third molars
* Systemic or infectious diseases that may impair wound healing, including active malignancy, diabetes mellitus with HbA1c > 7.0%, history of head and neck radiotherapy, true xerostomia, and HIV/AIDS
* Cervical caries, non-carious cervical lesions, or Class V restorations interfering with the CEJ
* Active periodontitis
* Use of medications affecting periodontal tissues or wound healing, including systemic corticosteroids, immunosuppressants, isotretinoin, bisphosphonates, and monoclonal antibodies with immunosuppressive, antiresorptive, or antiangiogenic effects
* Smoking
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Mean Root Coverage (MRC, %) | 6 months and 12 months post-surgery
  Mean root coverage (MRC), expressed as a percentage (%), assessed at 6 and 12 months post-surgery.
  MRC is calculated as (GR₀ - GR₆) / GR₀ × 100% and (GR₀ - GR₁₂) / GR₀ × 100%, respectively.
  Gingival recession (GR), measured in millimeters (mm) as the distance from the cemento-enamel junction (CEJ) to the gingival margin at the mid-buccal aspect of the tooth, is used solely as an input parameter for the calculation of MRC.

SECONDARY OUTCOMES:
Gingival recession height (GRH, mm) | baseline, 6 months, and 12 months post-surgery
  Distance from the cemento-enamel junction (CEJ) to the gingival margin measured at the mid-buccal aspect of the tooth.
Gingival recession width (RW, mm) | baseline, 6 months, and 12 months post-surgery
  Horizontal distance measured at the level of the cemento-enamel junction (CEJ) between the mesial and distal margins of the gingival recession.
Clinical Attachment Level (CAL, mm) | Baseline; 6 and 12 months post-surgery
  Distance from the cemento-enamel junction (CEJ) to the bottom of the gingival sulcus.
Probing Pocket Depth (PPD, mm) | baseline, 6 months, and 12 months post-surgery
  Distance from the gingival margin to the bottom of the gingival sulcus.
Gingival Thickness (GT, mm) | baseline, 6 months, and 12 months post-surgery
  Thickness of the gingiva measured 3 mm apical to the gingival margin at the mid-buccal aspect of the tooth.
Keratinized tissue width (KTW, mm) | baseline, 6 months, and 12 months post-surgery
  Distance from the gingival margin to the mucogingival junction
Complete Root Coverage (CRC, %) | 6 months and 12 months post-surgery
  % CRC = (number of teeth with CRC = 1 after treatment / total number of teeth with gingival recession at baseline) × 100.
  CRC = 1: postoperative GR ≤ 0 mm, indicating complete root coverage. CRC = 0: postoperative GR > 0 mm, indicating partial or no root coverage.
Gingival Recession Reduction (GR red, mm) | 6 months and 12 months post-surgery
  Reduction in recession height at 6 months: GR₀ - GR₆ Reduction in recession height at 12 months: GR₀ - GR₁₂
Clinical Attachment Level Gain (CAL Gain, mm) | 6 months and 12 months post-surgery
  Clinical attachment level gain at 6 months = CAL₀ - CAL₆
  Clinical attachment level gain at 12 months = CAL₀ - CAL₁₂
Keratinized Tissue Width Gain (KTW Gain, mm) | 6 months and 12 months post-surgery
  Increase in keratinized tissue width at 6 months: KTW₆ - KTW₀ Increase in keratinized tissue width at 12 months: KTW₁₂ - KTW₀
Tooth Sensitivity (SEN, Schiff score) | Assessed on the day of surgery before administration of anesthesia, and subsequently at 6 and 12 months after surgery.
  Clinician-assessed tooth sensitivity evaluated using the Schiff Cold Air Sensitivity Scale.
  Air will be delivered using a standard air syringe of the dental unit, positioned approximately 1 cm from the tooth surface for 5 seconds, at a working temperature of 23 °C (±4 °C), and directed at the exposed buccal surface of the tooth with gingival recession.
  Patient response to the air stimulus will be assessed by the clinician using the Schiff Cold Air Sensitivity Scale as follows:
  0 = No response to the air stimulus
  1. = Response to the air stimulus, but no request to discontinue the stimulus
  2. = Response to the air stimulus, with a request to discontinue the stimulus and/or turning away from the stimulus
  3. = Painful response to the air stimulus, with a request to discontinue the stimulus
Root Esthetic Score (RES, score) | 6 and 12 months after surgery
  Root Esthetic Score (RES), expressed as a composite score ranging from 0 to 10 points.
  The RES is a clinician-assessed composite esthetic outcome comprising the following five components:
  1. Gingival Margin (GM): failure of root coverage (0 points), partial root coverage (3 points), complete root coverage (6 points);
  2. Marginal Tissue Contour (MTC): irregular gingival margin not following the cemento-enamel junction (CEJ) (0 points), scalloped gingival contour following the CEJ (1 point);
  3. Soft Tissue Texture (STT): presence of scar (0 points), absence of scars (1 point);
  4. Mucogingival Junction (MGJ): MGJ not aligned with the MGJ of adjacent teeth (0 points), MGJ aligned with the MGJ of adjacent teeth (1 point);
  5. Gingival Color (GC): color mismatch with adjacent teeth (0 points), color matching adjacent teeth (1 point).
  The total RES score is calculated as the sum of all component scores, with higher scores indicating a better esthetic outcome.
Discomfort during the procedure (VAS, 0-10) | Immediately after completion of the procedure
  Patient-reported discomfort during the procedure assessed using the Visual Analogue Scale (VAS; 0 = no discomfort, 10 = extreme discomfort).
Pain intensity (VAS scale, 0-10) | 1, 2, 4, 7, 14 days after procedure
  Patient-reported pain intensity assessed using the Visual Analogue Scale (VAS; 0 = no pain, 10 = maximum pain).
Postoperative swelling (VAS scale, 0-10) | 1, 2, 4, 7, 14 days after procedure
  Patient-reported swelling assessed using the Visual Analogue Scale (VAS; 0 = none, 10 = maximum).
Tooth sensitivity (VAS, 0-10) | 1, 2, 4, 7, and 14 days post-procedure
  Patient-reported tooth sensitivity assessed using the Visual Analogue Scale (VAS; 0 = none, 10 = maximum).
Gingival color (VAS, 0-10) | 6 and 12 months post-surgery
  Patient-reported gingival color assessed using the Visual Analogue Scale (VAS; 0 = very poor, 10 = excellent).
Gingival shape (VAS 0-10) | 6 and 12 months post-surgery
  Patient-reported gingival shape assessed using a single Visual Analogue Scale (VAS; 0 = very poor, 10 = excellent)
Tooth appearance (VAS, 0-10) | 6 and 12 months post-surgery
  Patient-reported tooth appearance assessed using the Visual Analogue Scale (VAS; 0 = very poor, 10 = excellent).

OTHER OUTCOMES:
Procedure-related stress (VAS, 0-10) | Baseline (day of surgery, pre-anesthesia)
  Patient-reported procedure-related stress assessed using the Visual Analogue Scale (VAS; 0 = no stress, 10 = extreme stress).
Treatment satisfaction (VAS, 0-10) | 12 months after surgery
  Patient-reported treatment satisfaction assessed using the Visual Analogue Scale (VAS; 0 = not satisfied at all, 10 = completely satisfied).
Willingness to choose the treatment again (yes/no) | 12 months after surgery
  Patient-reported willingness to choose the same treatment again assessed using a dichotomous (yes/no) question.
Willingness to recommend the treatment (yes/no) | 12 months after surgery
  Patient-reported willingness to recommend the treatment to others assessed using a dichotomous (yes/no) question.

CONTACTS AND LOCATIONS:
Overall Officials: Bartłomiej Górski, Study Chair — Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw, Warsaw, Mazowsze, Poland